CLINICAL TRIAL: NCT01809613
Title: Functional Magnetic Resonance Imaging (fMRI) During Deep Brain Stimulation (DBS) to Treat Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kendall H. Lee, PI, Mayo Clinic
Other Study IDs: 12-009020
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Parkinson Disease; Essential Tremor; Dystonia; Obsessive Compulsive Disorder
Keywords: Parkinson disease; Deep Brain Stimulation; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deep Brain Stimulation: Functional Magnetic Resonance Imaging (fMRI) will be performed to determine the areas of BOLD signal modulation with DBS.
  Interventions: Procedure: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Procedure: Functional Magnetic Resonance Imaging (fMRI) — During the deep brain stimulation (DBS) surgery of the subthalamic nucleus within the thalamocortical basal ganglion, an additional lead extendor will be connected to the DBS electrode to allow externalization of the lead. Following confirmation of electrode location with MRI, a series of fMRI scans will be run. Total scanning time will be limited to 35 minutes.

SUMMARY:
This study is investigating the usefulness of using functional magnetic resonance imaging (fMRI) to monitor brain activation during deep brain stimulation for Parkinson's Disease, Essential tremor, dystonia, OCD, depression, pain, Tourette's syndrome, and epilepsy. The study may determine the relationship between patterns of brain activation and therapeutic outcome and/or side effects.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an effective neurosurgical approach for treating motor disorders including Parkinson's disease (PD), Essential Tremor (ET), and dystonia. Its therapeutic benefit has led to the application of DBS to a wide spectrum of disorders including psychiatric conditions, epilepsy, Alzeimer's disease, headache, obsessive-compulsive disorder (OCD), Tourette syndrome, depression and intractable pain. However, because the nature of its underlying mechanisms and clinical effects are not fully understood, precision targeting, decreasing adverse effects, and improving clinical outcomes represent major clinical and scientific challenges in PD and other disorders treated by DBS. Our goal is to investigate the inter-relationships between site-specific neural activation and clinical outcomes during DBS. To do so, we will perform non-invasive functional Magnetic Resonance Imaging (fMRI) to investigate DBS-mediated activation of neural network circuitry. Our proposed protocol involves the addition of intraoperative fMRI to the standard DBS or battery change protocol in order to determine the major sites of activation during application of clinically effective DBS to the subthalamic nucleus (STN), ventral intermediate thalamus (VIM), globus pallidus interna (GPi), fornix, nucleus accumbens (NAc), anterior thalamus and periaqueductal gray matter. Patients will undergo clinical assessment to determine the relative efficacy of DBS stimulation parameters, applied during the fMRI and at regularly scheduled post-operative programming visits up to 6 months of follow-up. Our Specific Aims are to: (1) Identify fMRI-activated brain regions by DBS in patients who undergo DBS surgery (Patients diagnosed with PD, ET, dystonia, OCD, depression, pain, Tourette's syndrome, and epilepsy. (2) Correlate fMRI activation with clinical outcomes and side effects. With the goal of improving DBS electrode targeting for optimal and reproducible clinical outcomes, these experiments will be the first attempt to relate site-specific DBS with functional in vivo imaging data and quantitative longitudinal clinical outcome measures in DBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients with medically intractable Parkinson's Disease who have been approved for DBS surgery by the interdisciplinary Mayo DBS committee.

Exclusion Criteria:

* Pregnant patients, prisoners, children (age less than 18), and any patients identified as unsuitable for this protocol by the Mayo DBS committee.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients approved and scheduled to undergo the clinical procedure of Deep Brain stimulation.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2013-03; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

PRIMARY OUTCOMES:
Mean Score on Unified Parkinson's Disease Rating Scale (UPDRS) | 6 months after Deep Brain Stimulation
  The UPDRS is a rating scale used to follow the longitudinal course of Parkinson's disease. The version of the scale used in this study has a total of 14 items; each of these item has a scale of 0-4, with 0 being no impairment, and 4 being severe impairment. All of the parts are combined to give a numeric score: 0 indicating no sign of disease, and 56, the highest score indicating severely incapacitated.

CONTACTS AND LOCATIONS:
Overall Officials: Kendall Lee, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Knight EJ, Testini P, Min HK, Gibson WS, Gorny KR, Favazza CP, Felmlee JP, Kim I, Welker KM, Clayton DA, Klassen BT, Chang SY, Lee KH. Motor and Nonmotor Circuitry Activation Induced by Subthalamic Nucleus Deep Brain Stimulation in Patients With Parkinson Disease: Intraoperative Functional Magnetic Resonance Imaging for Deep Brain Stimulation. Mayo Clin Proc. 2015 Jun;90(6):773-85. doi: 10.1016/j.mayocp.2015.03.022. PMID 26046412